CLINICAL TRIAL: NCT02796664
Title: Preventive Effects of Ginseng Against Atherosclerosis and Subsequent Ischemic Stroke: A Randomized Controlled Trial
Brief Title: Preventive Effects of Ginseng Against Atherosclerosis
Acronym: PEGASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dae Chul Suh (Other)
Collaborators: Korea Ginseng Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dae Chul Suh, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KGC2016-26
Record Dates: First submitted 2016-05-26; First posted 2016-06-13 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke; Atherosclerosis
Keywords: Ginseng; Stroke; Quantitative magnetic resonance flow analysis
MeSH Terms: conditions — Ischemic Stroke; Atherosclerosis; Stroke | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginseng (Experimental)
  Interventions: Dietary Supplement: Ginseng
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginseng — Korean Red Ginseng extract tablet (0.5 grams/tablet, 2 tablets twice a day) daily for 12 months.
  Arms: Ginseng
Dietary Supplement: Placebo — Placebo (0.5 grams/tablet, 2 tablets twice a day) daily for 12 months.
  Arms: Placebo

SUMMARY:
This study is a 12-month, double-blind, randomized, placebo-controlled trial. The purpose of this study is to determine whether ginseng is effective in the prevention of atherosclerosis and subsequent ischemic stroke. High-risk patients with severe atherosclerosis in the major intracranial arteries and extracranial carotid artery were enrolled.

ELIGIBILITY:
"Inclusion Criteria"

Patients were included if they

1. were aged 20 to 80 years;
2. had occlusion or severe stenosis (≥ 70%) of extracranial carotid artery and major intracranial arteries (intracranial carotid artery, middle cerebral artery, anterior cerebral artery, intracranial vertebral, basilar, or posterior cerebral artery) as documented by cerebral catheter angiography;
3. had any risk factor for stroke, such as hypertension, diabetes mellitus, hypercholesterolemia, smoking, alcohol drinking, or previous stroke history;
4. had no adverse reactions to administration of ginseng; and
5. agreed to participate in the trial.

"Exclusion Criteria"

Patients were excluded if they

1. did not agree to participate in the trial;
2. had any genetic cerebrovascular diseases;
3. had adverse reactions to contrast medium;
4. were pregnant or planning to be pregnant;
5. had a history of cardioembolic stroke;
6. had an emboligenic cardiac disease such as atrial fibrillation, valve disease, congestive heart failure, or recent myocardial infarction;
7. had a risk of stroke of other determined etiology according to the TOAST classification;
8. had undergone any neurointervention procedure or surgery, such as intra-arterial thrombolysis, angioplasty procedures, carotid endarterectomy, or bypass surgery;
9. had chronic kidney disease (GFR < 30 ml/min); or
10. had severe hepatic dysfunction.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dae Chul Suh, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng M, Xin Y, Li Y, Xu F, Xi X, Guo H, Cui X, Cao H, Zhang X, Han C. Ginsenosides: A Potential Neuroprotective Agent. Biomed Res Int. 2018 May 8;2018:8174345. doi: 10.1155/2018/8174345. eCollection 2018. PMID 29854792
- [Background] Zhou Y, Li HQ, Lu L, Fu DL, Liu AJ, Li JH, Zheng GQ. Ginsenoside Rg1 provides neuroprotection against blood brain barrier disruption and neurological injury in a rat model of cerebral ischemia/reperfusion through downregulation of aquaporin 4 expression. Phytomedicine. 2014 Jun 15;21(7):998-1003. doi: 10.1016/j.phymed.2013.12.005. Epub 2014 Jan 22. PMID 24462216
- [Background] Bao C, Wang Y, Min H, Zhang M, Du X, Han R, Liu X. Combination of ginsenoside Rg1 and bone marrow mesenchymal stem cell transplantation in the treatment of cerebral ischemia reperfusion injury in rats. Cell Physiol Biochem. 2015;37(3):901-10. doi: 10.1159/000430217. Epub 2015 Sep 18. PMID 26384017
- [Background] Aleshin S, Strokin M, Sergeeva M, Reiser G. Peroxisome proliferator-activated receptor (PPAR)beta/delta, a possible nexus of PPARalpha- and PPARgamma-dependent molecular pathways in neurodegenerative diseases: Review and novel hypotheses. Neurochem Int. 2013 Oct;63(4):322-30. doi: 10.1016/j.neuint.2013.06.012. Epub 2013 Jun 25. PMID 23811400
- [Background] Kernan WN, Viscoli CM, Furie KL, Young LH, Inzucchi SE, Gorman M, Guarino PD, Lovejoy AM, Peduzzi PN, Conwit R, Brass LM, Schwartz GG, Adams HP Jr, Berger L, Carolei A, Clark W, Coull B, Ford GA, Kleindorfer D, O'Leary JR, Parsons MW, Ringleb P, Sen S, Spence JD, Tanne D, Wang D, Winder TR; IRIS Trial Investigators. Pioglitazone after Ischemic Stroke or Transient Ischemic Attack. N Engl J Med. 2016 Apr 7;374(14):1321-31. doi: 10.1056/NEJMoa1506930. Epub 2016 Feb 17. PMID 26886418
- [Background] Yang Y, Li X, Zhang L, Liu L, Jing G, Cai H. Ginsenoside Rg1 suppressed inflammation and neuron apoptosis by activating PPARgamma/HO-1 in hippocampus in rat model of cerebral ischemia-reperfusion injury. Int J Clin Exp Pathol. 2015 Mar 1;8(3):2484-94. eCollection 2015. PMID 26045754
- [Background] Liu XY, Zhou XY, Hou JC, Zhu H, Wang Z, Liu JX, Zheng YQ. Ginsenoside Rd promotes neurogenesis in rat brain after transient focal cerebral ischemia via activation of PI3K/Akt pathway. Acta Pharmacol Sin. 2015 Apr;36(4):421-8. doi: 10.1038/aps.2014.156. Epub 2015 Mar 16. PMID 25832422
- [Background] Chen LM, Zhou XM, Cao YL, Hu WX. Neuroprotection of ginsenoside Re in cerebral ischemia-reperfusion injury in rats. J Asian Nat Prod Res. 2008 May-Jun;10(5-6):439-45. doi: 10.1080/10286020801892292. PMID 18464084
- [Background] He B, Chen P, Yang J, Yun Y, Zhang X, Yang R, Shen Z. Neuroprotective effect of 20(R)-ginsenoside Rg(3) against transient focal cerebral ischemia in rats. Neurosci Lett. 2012 Sep 27;526(2):106-11. doi: 10.1016/j.neulet.2012.08.022. Epub 2012 Aug 19. PMID 22925661
- [Background] Hong KS. Blood Pressure Management for Stroke Prevention and in Acute Stroke. J Stroke. 2017 May;19(2):152-165. doi: 10.5853/jos.2017.00164. Epub 2017 May 31. PMID 28592775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in a single center, from June 2016 to June 2017.
Period: Overall Study
Arm/Group | Ginseng | Placebo
Started | 29 | 29
Completed | 28 | 24
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Noncompliance | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ginseng | Placebo | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.5) | 58.8 (13.6) | 60.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 28 | 24 | 52
Hypertension [Count of Participants; unit: Participants] | 20 | 14 | 34
Diabetes mellitus [Count of Participants; unit: Participants] | 10 | 4 | 14
Hyperlipidemia [Count of Participants; unit: Participants] | 23 | 15 | 38
Previous stroke history [Count of Participants; unit: Participants] | 13 | 9 | 22
Atrial fibrillation [Count of Participants; unit: Participants] | 0 | 0 | 0
Myocardial infarction [Count of Participants; unit: Participants] | 0 | 0 | 0
Angina pectoris [Count of Participants; unit: Participants] | 5 | 2 | 7
Alcohol drinking [Count of Participants; unit: Participants] | 6 | 9 | 15
Smoking [Count of Participants; unit: Participants] | 5 | 13 | 18
Antiplatelet medication [Count of Participants; unit: Participants]
  Mono antiplatelet | 8 | 9 | 17
  Dual antiplatelet | 17 | 14 | 31
  Other antiplatelet | 2 | 1 | 3
  None | 1 | 0 | 1
Antihypertensive medication [Count of Participants; unit: Participants] | 21 | 13 | 34
Antidiabetic medication [Count of Participants; unit: Participants] | 9 | 3 | 12
Antihyperlipidemic medication [Count of Participants; unit: Participants] | 25 | 21 | 46
Baseline modified Rankin Scale (mRS) [Count of Participants; unit: Participants] — The modified Rankin scale (mRS) is a 6 point disability scale with possible scales ranging from 0 to 5. If the patient has no stroke symptoms, the value of the mRS is 0; able to carry out all pre-stroke activities, 1; unable to carry out all pre-stroke activities but is able to look after self without daily help, 2; requires some external help but is able to walk without the assistance of another individual, 3; unable to walk or attend to bodily functions without the assistance of another individual, 4; bedridden, incontinent, requires continuous care, 5.
  Participants
    mRS 0 | 21 | 22 | 43
    mRS 1 | 5 | 1 | 6
    mRS 2 | 0 | 0 | 0
    mRS 3 | 2 | 1 | 3
    mRS 4 | 0 | 0 | 0
    mRS 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Composite of Cerebral Ischemic Stroke and Transient Ischemic Attack
Description: The 1-year composite of cerebral ischemic stroke and transient ischemic attack downstream to an atherosclerotic lesion
Time Frame: Twelve months after randomization.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
Participants
  Ischemic stroke | 0 | 0
  Transient ischemic attack | 0 | 1
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and cerebral ischemic events including ischemic stroke and transient ischemic attack. The number of participants who suffered ischemic stroke and the number of paticipants who suffered transient ischemic attack were analyzed together to test the null hypothesis in two by two table; Test type: Other — Equality test; p = 0.462, Fisher Exact

2. Primary Outcome: Modified Rankin Scale
Description: Presence of other cerebro-cardiovascular morbidity or mortality assessed by aggravation of patient status (modified Rankin Scale). The modified Rankin Scale is ranging from 0 to 5. The higher scale indicates the worse outcome.
Time Frame: Twelve months after randomization.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
Participants
  mRS 0 | 21 | 22
  mRS 1 | 5 | 1
  mRS 2 | 0 | 0
  mRS 3 | 2 | 1
  mRS 4 | 0 | 0
  mRS 5 | 0 | 0
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and modified Rankin Scale at follow-up; Test type: Other — Equality test; p = 0.34, Fisher Exact

3. Secondary Outcome: The Changes in Volumetric Blood Flow (ml/Sec) in Intracranial Vessels.
Description: The changes in volumetric blood flow (ml/sec) in intracranial vessels assessed by quantitative magnetic resonance angiography with noninvasive optimal vessel analysis.
Time Frame: At randomization and twelve months after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
Participants
  The flow change in steno-occlusive lesion: Improved | 4 | 5
  The flow change in steno-occlusive lesion: No change | 17 | 18
  The flow change in steno-occlusive lesion: Aggravated | 7 | 1
  The flow change in collateral vessel: Improved | 7 | 7
  The flow change in collateral vessel: No change | 17 | 9
  The flow change in collateral vessel: Aggravated | 4 | 8
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and flow change in steno-occlusive lesion; Test type: Other — Equality test; p = 0.13, Fisher Exact
Statistical Analysis 2: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and flow change in collateral vessel; Test type: Other — Equality test; p = 0.17, Chi-squared

4. Secondary Outcome: The Changes of White Matter Hyperintensities.
Description: The changes of white matter hyperintensities, assessed by the Fazekas scale using brain magnetic resonance imaging. The Fazekas scale is a 4 point white matter disease severity scale with values ranging from 0 to 3. It quantifies the amount of white matter T2 hyperintense lesions each in periventricular white matter and deep white matter. Higher scales mean a worse white matter status. In the region of the periventricular white matter, 0 means absence of the lesion; 1, caps or pencil-thin lining lesion; 2, smooth halo lesion; 3, irregular high intense signal extending into the deep shite matter. In the region of the deep white matter, 0 means absence of the lesion; 1, punctate foci lesions; 2, beginning confluence; 3, large confluent hyperintense areas.
Time Frame: At randomization and twelve months after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
Participants
  Periventricular white matter: Fazekas scale 0 | 2 | 1
  Periventricular white matter: Fazekas scale 1 | 9 | 11
  Periventricular white matter: Fazekas scale 2 | 15 | 10
  Periventricular white matter: Fazekas scale 3 | 2 | 2
  Deep white matter: Fazekas scale 0 | 9 | 6
  Deep white matter: Fazekas scale 1 | 15 | 15
  Deep white matter: Fazekas scale 2 | 3 | 2
  Deep white matter: Fazekas scale 3 | 1 | 1
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and periventricular white matter lesions at follow-up; Test type: Other — Equality test; p = 0.74, Fisher Exact
Statistical Analysis 2: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and deep white matter lesions at follow-up; Test type: Other — Equality test; p = 0.95, Fisher Exact

5. Secondary Outcome: Number of Participants With Changes of Parenchymal Ischemic Lesions
Description: The changes of ischemic parenchymal lesions, assessed by brain magnetic resonance images acquired at randomization and twelve months after randomization. We counted the number of participants who had new ischemic parenchymal lesions at twelve months after randomization.
Time Frame: At randomization and twelve months after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
Participants
  Ischemic lesion (+) | 22 | 15
  Ischemic lesion (-) | 6 | 9
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and parenchymal ischemic lesions at follow-up; Test type: Other — Equality test; p = 0.23, Chi-squared

6. Other Pre Specified Outcome: Drug Compliance
Description: We calculated average drug compliance based on the number of remained drugs at each follow-up.
Time Frame: At twelve months after randomization.
Measure: Mean (Standard Deviation); unit: percentage of drug compliance
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 28 | 24
percentage of drug compliance | 97.4 (4.7) | 97.8 (4.3)
Statistical Analysis 1: Comparison: Ginseng vs Placebo; The null hypothesis is that there is no relationship between ginseng administration and drug compliance at follow-up; Test type: Other — Equality test; p = 0.79, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1, 3, 6 and 12 months after randomization.
Arm/Group | Ginseng | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/29
Other Adverse Events (participants affected / at risk) | 1/29 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginseng (N=29) | Placebo (N=29)
Death (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginseng (N=29) | Placebo (N=29)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subjective hair loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1. The difficulty in determining the size of the study population due to the lack of previous studies.
2. The relatively short follow-up period considering chronic atherosclerotic disease.
3. The absence of surrogate biochemical markers to confirm ginsenosides' effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02796664/Prot_SAP_000.pdf